CLINICAL TRIAL: NCT05011695
Title: Comparison of the Effectiveness of Different Treatment Methods in Patients With Plantar Fasciitis
Brief Title: Different Treatment Methods in Patients With Plantar Fasciitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Seyit Çıtaker, Prof.Dr., Gazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HRU/21.10.21
Record Dates: First submitted 2021-08-10; First posted 2021-08-18 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-08

CONDITIONS: Plantar Fasciitis
Keywords: Plantar fasciitis; exercise; ESWT; physical therapy
MeSH Terms: conditions — Fasciitis, Plantar; Motor Activity | interventions — Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: Patients will be divided into 3 groups. The 1st group will be given ESWT therapy, the 2nd group will be given transverse friction massage, and the 3rd group will be given exercises that are used in the treatment of plantar fasciitis and have proven effectiveness.
Who Masked: Participant
Masking Description: Patients will not know which treatment group they are in.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 1. Group ESWT treatment (Active Comparator): 6000 SWT Easy" device will be used for ESWT treatment. The plantar fascia of the patients will be applied once a week for 3 weeks. In each application, 2400 beats, 2.0 bar pressure and 12 frequency doses of ESWT will be applied
  Interventions: Other: physiotherapy
- 2. Group transverse friction massage (Active Comparator): Transverse friction massage will be applied to the plantar fascia of the patients for 3 weeks, 3 days a week, on Mondays, Wednesdays, and Fridays, with a break for 1 day and 15 minutes each. Transverse friction massage, when the patient is in the supine semi-lying position, the big toe will be dorsiflexed and in this position, it will be applied in the direction that will be transverse to the plantar fascia.
  Interventions: Other: physiotherapy
- 3. Group exercise group (Active Comparator): Stretching the plantar fascia and gastrocsoleus muscles of the patients, towel picking exercises with the foot intrinsic muscles, heel drop exercises will be given. All stretching and exercises will be applied once a day, 5 days a week, for 3 weeks. Plantar fascia stretching exercises will be performed with a physiotherapist; While the patient is lying in the supine position, 30 seconds of stretching will be performed using the windlass (windlass) mechanism (toes are brought to dorsi flexion). This stretch will be repeated 3 times. Gastrocsoleus stretching exercises will be studied with a physiotherapist. In the supine position, the gastrocsoleus muscles will be stretched for 10 seconds and stretching will be performed with 10 repetitions. Towel collection exercises for the foot intrinsic muscles will be practiced in 3 sets, 15 repetitions per day. Heel drop exercise will be applied in 3 sets of 15 repetitions per day.
  Interventions: Other: physiotherapy

INTERVENTIONS:
Other: physiotherapy — The 1st group will be given ESWT therapy, the 2nd group will be given transverse friction massage, and the 3rd group will be given exercises that are used in the treatment of plantar fasciitis and have proven effectiveness

SUMMARY:
The aim of this study is to determine the different treatment methods efficacy in adult individuals with plantar fasciitis. Pain, functionality level, range of motion, muscle performance, quality of life will be examined.

In the studies carried out to date; The comparison of the effectiveness of stretching exercises and Extracorporeal shock wave therapy (ESWT), the comparison of ESWT therapy and ultrasound therapy, the comparison of manual therapy methods and stretching exercises were studied. The effects of the use of double air cushion shoes and exercise therapy on pain management and functional status were investigated.

However, no study has been conducted to compare the effectiveness of ESWT treatment, transverse friction massage and exercise training, and to determine whether technics have superiority over each other. In this study, in addition to the evaluation of pain and functionality; joint range of motion, muscle performance and quality of life are the distinguishing features of the study. That's why researcher came up with the idea to work on this topic. This study will shed light on future studies and will contribute to the literature in the treatment of this diagnosis group. It will give us information about whether the different treatment methods researcher use in physical therapy are superior to each other.

DETAILED DESCRIPTION:
This study will be conducted with adults over the age of 18, who applied to the Şanlıurfa Training and Research Hospital Physical Therapy Unit, were diagnosed with plantar fasciitis, had pain for at least 3 months, and agreed to participate in the study. Patients with diabetes, systemic inflammatory disease, previous foot injury, foot fracture or malignancy, neurological disease and pregnant women will not be included in the study. A total of 54 people will be included in the study. Patients will be divided into 3 groups of 18 people each in a randomized controlled manner with a computer program. Different treatment methods with proven effectiveness in the treatment of plantar fasciitis will be applied to each group. The 1st group will be given ESWT therapy, the 2nd group will be given transverse friction massage, and the 3rd group will be given exercises that are used in the treatment of plantar fasciitis and have proven effectiveness.

1. Group ESWT treatment: "6000 SWT Easy" device will be used for ESWT treatment. The plantar fascia of the patients will be applied once a week for 3 weeks. In each application, 2400 beats, 2.0 bar pressure and 12 frequency doses of ESWT will be applied.
2. Group transverse friction massage: Transverse friction massage will be applied to the plantar fascia of the patients for 3 weeks, 3 days a week, on Mondays, Wednesdays, and Fridays, with a break for 1 day and 15 minutes each. Transverse friction massage, when the patient is in the supine semi-lying position, the big toe will be dorsiflexed and the plantar fascia will be stretched, and in this position, it will be applied in the direction that will be transverse to the plantar fascia.
3. Group exercise group: Stretching the plantar fascia and gastrocsoleus muscles of the patients, towel picking exercises with the foot intrinsic muscles, heel drop exercises will be given. All stretching and exercises will be applied once a day, 5 days a week, for 3 weeks. Plantar fascia stretching exercises will be performed with a physiotherapist; While the patient is lying in the supine position, 30 seconds of stretching will be performed using the windlass (windlass) mechanism (toes are brought to dorsi flexion). This stretch will be repeated 3 times. Gastrocsoleus stretching exercises will be studied with a physiotherapist. In the supine position, the gastrocsoleus muscles will be stretched for 10 seconds and stretching will be performed with 10 repetitions. Towel collection exercises for the foot intrinsic muscles will be practiced in 3 sets, 15 repetitions per day. Heel drop exercise will be applied in 3 sets of 15 repetitions per day.

All patients will be evaluated before treatment and 3 days after the end of 3 weeks of treatment. In the evaluations to be made; Sociodemographic information such as diagnosis, age, height, weight, education level, gender of the patients will be recorded with the prepared data registration form.

Pain sensation will be evaluated with a visual analog scale. For pain severity, a 100mm horizontal line will be written as 0 points at the beginning "no pain" and 10 points at the end of "worst pain imaginable". Patients will be asked to mark the pain patients feel on this 100 mm long horizontal line. The length of the place marked by the patient will be recorded in mm. Pain at rest, during activity, and at night will be evaluated.

Foot functional evaluation will be done with the foot function index. This index consists of 3 sub-scales in which various functional states and pain sensation are evaluated and a total of 23 questions. Patients will score the questions in these subscales between 0 and 10. It will be evaluated out of 230 points in total. The higher the score, the worse the functional status is affected.

Functional status will be evaluated with triple hop test. The patient will be asked to stand on a single extremity to be tested and hop forward 3 times consecutively at the maximum level, the total distance taken will be recorded, the average of the 3 repetitions will be taken and recorded in cm.

Joint range of motion will be evaluated with a universal goniometer. The patient will be asked to bring the ankle to dorsi flexion and plantar flexion while lying on back, and how far patient can move will be measured in degrees with a goniometer. The active maximum amount of movement made by the patient will be measured and recorded in degrees (°).

Quality of life will be evaluated with the Short Form-36 scale. The scale consists of 8 sub-parameters and 36 questions. These sub-parameters are; physical function, body pain, limitation due to physical problems, limitation due to emotional problems, emotional well-being, social function, energy/fatigue, general health perception. The higher the score obtained from the scale, the higher the patient's quality of life.

The performance of the foot flexor muscles will be evaluated with the heel rise test. While standing, the patient will be asked to raise the heel as many times as possible for 30 seconds. How many times patients raise their heels in 30 seconds will be recorded.

For this study, permission was obtained from the Harran University Health Sciences Institute Non-Drug Clinical Research Ethics Committee before starting the research.

ELIGIBILITY:
Inclusion Criteria:

* unilateral plantar fasciitis
* adults over the age of 18
* diagnosis of plantar fasciitis
* pain for at least 3 months

Exclusion Criteria:

* diabetes
* systemic inflammatory disease
* previous foot injury
* foot fracture
* foot malignancy
* neurological disease
* pregnant women.
* Those who have received physical therapy before
* Those who have had prp before
* Those who have had a previous steroid injection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2021-06-11 (Actual); Primary Completion 2022-06-14 (Estimated); Study Completion 2022-12-19 (Estimated)

PRIMARY OUTCOMES:
Pain will be examined | three weeks
  Pain sensation will be evaluated with a visual analog scale. Patients can score a minimum of 0 and a maximum of 10. Getting a high score indicates a bad situation.

CONTACTS AND LOCATIONS:
Overall Officials: Seyit s ÇITAKER, Phd, Principal Investigator — Gazi University
Locations (1):
- Gazi University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
After the study is completed, its content will be shared with all researchers.

REFERENCES:
- [Result] Wheeler PC, Tattersall C. Extracorporeal Shockwave Therapy Plus Rehabilitation for Patients With Chronic Plantar Fasciitis Might Reduce Pain and Improve Function but Still Not Lead to Increased Activity: A Case-Series Study With Multiple Outcome Measures. J Foot Ankle Surg. 2018 Mar-Apr;57(2):339-345. doi: 10.1053/j.jfas.2017.07.001. Epub 2017 Oct 9. PMID 29032913
- [Result] Ugurlar M, Sonmez MM, Ugurlar OY, Adiyeke L, Yildirim H, Eren OT. Effectiveness of Four Different Treatment Modalities in the Treatment of Chronic Plantar Fasciitis During a 36-Month Follow-Up Period: A Randomized Controlled Trial. J Foot Ankle Surg. 2018 Sep-Oct;57(5):913-918. doi: 10.1053/j.jfas.2018.03.017. PMID 30149850
- See also: Pub med no 30149850 — https://pubmed.ncbi.nlm.nih.gov/30149850/
- See also: Pub med no 29032913 — https://pubmed.ncbi.nlm.nih.gov/29032913/